CLINICAL TRIAL: NCT02183259
Title: Absolute Bioavailability, Pharmacokinetics and Safety of ESR 1150 CL 1 mg Capsule Compared to 0.015 mg Solution i.v. as Single Administration in Healthy Male Subjects (Open-labelled, 2-way Cross-over Study)
Brief Title: Bioavailability, Pharmacokinetics and Safety of ESR 1150 CL in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1172.1
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Capsules; Solutions

ARMS (2):
- ESR 1150 CL capsule (Experimental)
  Interventions: Drug: ESR 1150 CL, Capsule, oral
- ESR 1150 CL ampoule (Experimental)
  Interventions: Drug: ESR 1150 CL, solution, intravenous

INTERVENTIONS:
Drug: ESR 1150 CL, Capsule, oral
  Arms: ESR 1150 CL capsule
Drug: ESR 1150 CL, solution, intravenous
  Arms: ESR 1150 CL ampoule

SUMMARY:
To investigate the bioavailability of ESR 1150 CL by the time course determination of plasma concentration (pharmacokinetics) of no-transformed ESR 1150 after single administration to healthy adult male volunteers. Secondary objective is to investigate the safety of ESR 1150 CL.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* age: >= 20 and <= 35 years
* weight: >= 50 to <= 80 kg and within +/- 20 % of standard weight
* blood pressure: systolic 100 - 138 mmHg and diastolic of less than 84 mmHg
* pulse rate: 45 to 80 beat/min
* volunteer whose participation in the trial is judged valid by the investigator based on the results of preliminary check-up and pre-administration check-up

Exclusion Criteria:

* history of diseases including cardiac, pulmonary, hepatic, renal or gastrointestinal disease
* history of drug allergy
* history of drug dependency, alcohol dependency, etc.
* use of other trial drug within 6 months before study drug administration
* use of any drugs within 7 days before study drug administration

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1998-11; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve from time zero to infinity | up to 16 hours after drug administration
maximum drug plasma concentration (Cmax) | up to 16 hours after drug administration
time to achieve maximum drug plasma concentration (tmax) | up to 16 hours after drug administration
elimination half-life (t1/2) | up to 16 hours after drug administration
mean residence time (MRT) | up to 16 hours after drug administration
total clearance (CL) | up to 16 hours after drug administration

SECONDARY OUTCOMES:
number of adverse events | up to day 22